CLINICAL TRIAL: NCT03624881
Title: Evaluation of the VISITAG SURPOINT™ Module With External Processing Unit (EPU) When Used With the THERMOCOOL SMARTTOUCH® SF and the THERMOCOOL SMARTTOUCH® Catheters for Pulmonary Vein Isolation (PVI) (SURPOINT COA)
Brief Title: Evaluation of VISITAG SURPOINT™ Module With External Processing Unit (EPU)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI_2017_06
Record Dates: First submitted 2018-07-26; First posted 2018-08-10 (Actual); Results first posted 2022-09-07 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- VISITAG SURPOINT Module with EPU (Experimental): Subjects undergoing electrophysiology mapping and RF ablation with THERMOCOOL SMARTTOUCH ® SF (STSF) and THERMOCOOL SMARTTOUCH ® (ST) catheters with VISITAG SURPOINT Module with External Processing Unit for pulmonary vein isolation
  Interventions: Device: Catheter ablation with EPU

INTERVENTIONS:
Device: Catheter ablation with EPU — Subjects undergoing electrophysiology mapping and RF ablation with THERMOCOOL SMARTTOUCH ® SF (STSF) and THERMOCOOL SMARTTOUCH ® (ST) catheters with VISITAG SURPOINT Module with External Processing Unit for pulmonary vein isolation

SUMMARY:
Prospective, non-randomized, post market clinical evaluation of the VISITAG SURPOINT™ Module with External Processing Unit (EPU) when used with STSF catheter and ST catheter compared to an historical control performance goal.

A maximum of 330 subjects will be enrolled across up to 45 sites. Two hundred eighty (280) enrolled subjects will be treated using the STSF catheter with EPU and 50 subjects will be treated using the ST catheter with EPU. Prior to enrollment, a few sites will be selected to only enroll subjects who will be treated with the ST catheter and the remaining sites will only enroll subjects who will be treated with the STSF catheter.

Bayesian adaptive design will be used to assess early success at up to two interims: one after all subjects have completed the 3- month follow-up assessment, and a second to occur after all subjects have completed the 6 months follow-up visit.

DETAILED DESCRIPTION:
Prospective, non-randomized, post market clinical evaluation of the VISITAG SURPOINT™ Module with External Processing Unit (EPU) when used with STSF catheter and ST catheter compared to an historical control performance goal.

A maximum of 330 subjects will be enrolled across up to 45 sites. Two hundred eighty (280) enrolled subjects will be treated using the STSF catheter with EPU and 50 subjects will be treated using the ST catheter with EPU. Prior to enrollment, a few sites will be selected to only enroll subjects who will be treated with the ST catheter and the remaining sites will only enroll subjects who will be treated with the STSF catheter.

Bayesian adaptive design will be used to assess early success at up to two interims: one after all subjects have completed the 3- month follow-up assessment, and a second to occur after all subjects have completed the 6 months follow-up visit.

The primary objective of this clinical investigation is to demonstrate the safety and 12-month effectiveness of Tag Index-guided ablation using the VISITAG SURPOINT™ Module with External Processing Unit when used with the THERMOCOOL SMARTTOUCH® SF (STSF) and THERMOCOOL SMARTTOUCH® (ST) catheters for pulmonary vein isolation (PVI) in the treatment of subjects with drug refractory symptomatic paroxysmal atrial fibrillation. Specifically:

* To demonstrate the safety based on the proportion of subjects with early-onset (within 7 days of ablation procedure) primary adverse events
* To demonstrate the 12-month effectiveness based on the proportion of subject with freedom from documented atrial arrhythmia (atrial fibrillation (AF), atrial tachycardia (AT) or atrial flutter (AFL) episodes during the effectiveness evaluation period (Day 91-365)

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Symptomatic paroxysmal AF who had at least one AF episode electrocardiographically documented within one (1) year prior to enrollment. Documentation may include electrocardiogram (ECG); Transtelephonic monitoring (TTM), Holter monitor or telemetry strip
2. Failed at least one antiarrhythmic drug (AAD) (Class I or III antiarrhythmic drugs) as evidenced by recurrent symptomatic AF, or intolerable to the AAD
3. Age 18 years or older
4. Signed Patient Informed Consent Form (ICF)
5. Able and willing to comply with all pre-, post-, and follow-up testing and requirements

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not eligible for enrollment.

1. Previous surgical or catheter ablation for atrial fibrillation
2. Previous cardiac surgery (including CABG) within the past 6 months (180 days)
3. Valvular cardiac surgical/percutaneous procedure (i.e., ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve)
4. Any carotid stenting or endarterectomy
5. Documented LA thrombus on imaging
6. LA size > 50 mm (parasternal long axis view)
7. LVEF < 40%
8. Contraindication to anticoagulation (heparin or warfarin)
9. History of blood clotting or bleeding abnormalities
10. PCI/MI within the past 2 months (60 days)
11. Documented thromboembolic event (including TIA) within the past 12 months (365 days)
12. Rheumatic Heart Disease
13. Uncontrolled heart failure or NYHA function class III or IV
14. Severe mitral regurgitation (Regurgitant volume ≥ 60 mL/beat, Regurgitant fraction ≥ 50%, and/or Effective regurgitant orifice area ≥ 0.40cm2)
15. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months (365 days)
16. Unstable angina
17. Acute illness or active systemic infection or sepsis
18. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
19. Presence of implanted ICD/CRT-D.
20. Significant pulmonary disease, (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms.
21. Gastroesophageal Reflux Disease (GERD; active requiring significant intervention not including OTC medication)
22. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
23. Women who are pregnant (as evidenced by pregnancy test if pre-menopausal)
24. Concurrent enrollment in an investigational study evaluating another device, biologic, or drug.
25. Presence of intracardiac thrombus, myxoma, tumor, interatrial baffle or patch or other abnormality that precludes vascular access, or manipulation of the catheter.
26. Life expectancy less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Grandview Medical Center, Birmingham, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - CHI St. Vincent, Little Rock, Arkansas
  - Scripps Health, San Diego, California
  - San Diego Cardiac Center, San Diego, California
  - Marian Regional Medical Center, Santa Maria, California
  - St. John's Providence, Santa Monica, California
  - University of Colorado Denver, Denver, Colorado
  - JFK Medical Center, Atlantis, Florida
  - Memorial Healthcare, Hollywood, Florida
  - Florida Hospital, Orlando, Florida
  - Baptist Hospital/Cardiology Consultants, Pensacola, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory St. Joseph's, Atlanta, Georgia
  - Evanston Community, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Prairie Heart Institute, Springfield, Illinois
  - Baptist Health Lexington, Kensington, Kentucky
  - Oschner LSU Health Shreveport, Shreveport, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Abbott Northwestern, Minneapolis, Minnesota
  - Lovelace Medical Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - NYU Langone, New York, New York
  - New York Presbyterian, New York, New York
  - Albert Einstein College of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Oklahoma Heart Institute, Oklahoma City, Oklahoma
  - Providence St Vincent Medical Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Erlanger Health System, Chattanooga, Tennessee
  - Texas Health Heart and Vascular Hospital, Arlington, Texas
  - St. David's Medical Center, Austin, Texas
  - Intermountain Medical, Murray, Utah
  - Sentara Health, Norfolk, Virginia
  - MultiCare Tacoma, Tacoma, Washington

REFERENCES:
- [Derived] Di Biase L, Monir G, Melby D, Tabereaux P, Natale A, Manyam H, Athill C, Delaughter C, Patel A, Gentlesk P, Liu C, Arkles J, McElderry HT Jr, Osorio J; SURPOINT Postapproval Trial Investigators. Composite Index Tagging for PVI in Paroxysmal AF: A Prospective, Multicenter Postapproval Study. JACC Clin Electrophysiol. 2022 Sep;8(9):1077-1089. doi: 10.1016/j.jacep.2022.06.007. Epub 2022 Aug 31. PMID 36137711

RESULTS

PARTICIPANT FLOW:
Groups:
- VISITAG SURPOINT Module STSF Catheter With EPU: Participants with symptomatic paroxysmal atrial fibrillation (PAF) who have failed at least one antiarrhythmic drug were treated with electrophysiology mapping and radiofrequency (RF) ablation using VISITAG SURPOINT module with THERMOCOOL SMARTTOUCH Surround Flow (STSF) catheter with external processing unit (EPU).
- VISITAG SURPOINT Module ST Catheter With EPU: Participants with symptomatic PAF who have failed at least one antiarrhythmic drug, were treated with electrophysiology mapping and radiofrequency (RF) ablation using VISITAG SURPOINT module with THERMOCOOL SMARTTOUCH (ST) catheter with EPU.
Period: Overall Study
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Started | 283 | 50
Safety Set | 261 | 49
Completed | 237 | 44
Not Completed | 46 | 6
Not completed — Screen Failure | 14 | 0
Not completed — No Catheter Inserted | 6 | 1
Not completed — Catheter Inserted and RF Energy Delivery with No EPU System Used | 2 | 0
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 10 | 4
Not completed — Withdrawal by Subject | 12 | 1

BASELINE CHARACTERISTICS:
Population: The safety set consisted of all enrolled participants who had undergone insertion of the STSF or ST catheter and use of the VISITAG SURPOINT module with EPU.
Groups:
- Total: Total of all reporting groups
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU | Total
Number analyzed (Participants) | 261 | 49 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (10.53) | 62.7 (9.97) | 63.4 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 27 | 136
  Male | 152 | 22 | 174
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 3 | 19
  Not Hispanic or Latino | 231 | 36 | 267
  Unknown or Not Reported | 14 | 10 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 11 | 0 | 11
  White | 221 | 37 | 258
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 24 | 9 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Primary Adverse Events (PAEs)
Description: A PAE is a serious adverse event (SAEs), which occurred within the first week (7 days) following an atrial fibrillation (AF) ablation procedure with use of Tag Index. Pulmonary vein (PV) stenosis and atrio-esophageal fistula that occurred greater than one week (7 days) post-procedure were deemed Primary AEs. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to 12 months
Population: The safety set consisted of all enrolled participants who had undergone insertion of the STSF or ST catheter and use of the VISITAG SURPOINT module with EPU. Here 'N' (number of participants analyzed) signifies the number of participants analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 261 | 48
Participants | 11 | 3

2. Primary Outcome: Number of Participants Free From Atrial Tachyarrhythmias (Symptomatic and Asymptomatic)
Description: Number of participants free from symptomatic and asymptomatic atrial tachyarrhythmias (which includes atrial fibrillation [AF], atrial flutter [AFL], and atrial tachycardia [AT]) were reported.
Time Frame: Up to 12 months
Population: The Per-protocol (PP) set consisted of all enrolled participants who had undergone RF ablation and were treated with the STSF or ST catheters with the VISITAG SURPOINT Module with EPU, and had been treated for the study-related arrhythmia. Here 'N' (number of participants analyzed) signifies the number of participants analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 228 | 44
Participants | 173 | 34

3. Secondary Outcome: Percentage of Participants With Cumulative PAEs
Description: A PAE is a serious adverse event, which occurs within the first week (7 days) following an AF ablation procedure with use of Tag Index. Pulmonary vein (PV) stenosis and atrio-esophageal fistula that occurs greater than one week (7 days) post-procedure were deemed Primary AEs. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to 12 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 261 | 49
Percentage of Participants | 4.3 | 6.3

4. Secondary Outcome: Number of Participants With Unanticipated Adverse Device Effects (UADEs)
Description: Number of participants with UADEs was reported.
Time Frame: Up to 12 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 261 | 49
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Serious Non-Primary AEs
Description: Serious non-primary adverse events were defined as serious AEs (SAEs) that are not primary adverse events. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to 12 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 261 | 49
Participants | 42 | 3

6. Secondary Outcome: Number of Participants With Bleeding Complication by International Society on Thrombosis and Haemostasis (ISTH) Class and Timing of Onset
Description: Number of participants with bleeding complication by ISTH class and timing of onset were reported. The ISTH classification of major bleeding event is a hemoglobin drop of greater than or equal to (>=) 2 grams per deciliter (g/dL), transfusion of >= 2 units (U) packed red blood cells, symptomatic bleed in a critical area, or fatal bleed. Clinically relevant non-major (CRNM) events require prolong hospitalization or result in laboratory testing, imaging, compression, procedure, interruption of the study medication or a change in concomitant therapy. Minor bleeding events are overt bleeding events that do not meet the criteria for CRNM or major bleeding events.
Time Frame: Within 7 Days (Early Onset), 8-30 Days (Peri-procedural) and >=31 Days (Late Onset) of Initial Ablation Procedure (Up to 12 Months)
Population: The safety set consisted of all enrolled participants who had undergone insertion of the STSF or ST catheter and use of the VISITAG SURPOINT module with EPU. Here 'n' (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 261 | 49
Participants
  Major (0-7 Days) | 0 | 0
  Major (8-30 Days): number analyzed (Participants) | 260 | 49
  Major (8-30 Days) | 0 | 0
  Major (>=31 Days): number analyzed (Participants) | 260 | 49
  Major (>=31 Days) | 0 | 0
  CRNM (0-7 Days) | 4 | 0
  CRNM (8-30 Days): number analyzed (Participants) | 260 | 49
  CRNM (8-30 Days) | 0 | 0
  CRNM (>=31 Days): number analyzed (Participants) | 260 | 49
  CRNM (>=31 Days) | 3 | 0
  Minor (0-7 Days) | 17 | 1
  Minor (8-30 Days): number analyzed (Participants) | 260 | 49
  Minor (8-30 Days) | 2 | 0
  Minor (>=31 Days): number analyzed (Participants) | 260 | 49
  Minor (>=31 Days) | 7 | 1

7. Secondary Outcome: Percentage of Participants With Ipsilateral Pulmonary Vein Isolation (PVI) (Entrance Block) at the End of the Procedure
Description: Percentage of participants with ipsilateral PVI (entrance block) at the end of the procedure were reported.
Time Frame: End of the Procedure (up to 12 months)
Population: The PP set consisted of all enrolled participants who had undergone RF ablation and were treated with the STSF or ST catheters with the VISITAG SURPOINT Module with EPU, and had been treated for the study-related arrhythmia.
Measure: Number; unit: Percentage of Participants
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 246 | 49
Percentage of Participants | 98.8 | 100

8. Secondary Outcome: Percentage of Participants With Ipsilateral PVI After First Encirclement Without Acute Reconnection
Description: Percentage of participants with ipsilateral PVI after first encirclement without Acute reconnection was reported.
Time Frame: Up to 12 months
Population: as for outcome 7
Measure: Number; unit: Percentage of Participants
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 246 | 49
Percentage of Participants | 72.0 | 85.7

9. Secondary Outcome: Percentage of Targeted Veins With Touch-up (Ablation of Acute Reconnection) Among All Targeted Veins
Description: Percentage of targeted veins with touch-up (ablation of acute reconnection) among all targeted veins was reported.
Time Frame: Up to 12 months
Population: as for outcome 7
Measure: Number; unit: Percentage of targeted veins
Units Other Than Participants: Targeted Veins
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 246 | 49
Number analyzed (Targeted Veins) | 492 | 98
Percentage of targeted veins | 16.9 | 7.1

10. Secondary Outcome: Percentage of Targeted Veins With Touch-up at Anatomical Location of Acute PV Reconnection After First Encirclement
Description: Percentage of targeted veins with touch-up at anatomical location of acute PV reconnection after first encirclement was reported. The location included anterior, superior, ridge, posterior, and inferior region of the left pulmonary veins (LPV) and right pulmonary veins (RPV).
Time Frame: Up to 12 months
Population: The PP set consisted of all enrolled participants who had undergone RF ablation and were treated with the STSF or ST catheters with the VISITAG SURPOINT Module with EPU, and had been treated for the study-related arrhythmia. Here 'n' (number of targeted veins analyzed) included all evaluable numbers of targeted veins which were analyzed at specified categories.
Measure: Number; unit: Percentage of targeted veins
Units Other Than Participants: Targeted Veins
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 246 | 49
Number analyzed (Targeted Veins) | 242 | 49
Percentage of targeted veins
  LPV: Anterior: number analyzed (Targeted Veins) | 166 | 41
  LPV: Anterior | 4.2 | 2.4
  LPV: Superior: number analyzed (Targeted Veins) | 173 | 32
  LPV: Superior | 3.5 | 0.0
  LPV: Ridge: number analyzed (Targeted Veins) | 230 | 45
  LPV: Ridge | 3.9 | 0.0
  LPV: Posterior: number analyzed (Targeted Veins) | 241 | 49
  LPV: Posterior | 7.5 | 0.0
  LPV: Inferior: number analyzed (Targeted Veins) | 238 | 46
  LPV: Inferior | 1.3 | 2.2
  RPV: Anterior: number analyzed (Targeted Veins) | 242 | 46
  RPV: Anterior | 11.6 | 4.3
  RPV: Superior: number analyzed (Targeted Veins) | 176 | 32
  RPV: Superior | 5.7 | 12.5
  RPV: Ridge: number analyzed (Targeted Veins) | 11 | 3
  RPV: Ridge | 9.1 | 0.0
  RPV: Posterior: number analyzed (Targeted Veins) | 241 | 49
  RPV: Posterior | 13.3 | 6.1
  RPV: Inferior: number analyzed (Targeted Veins) | 237 | 47
  RPV: Inferior | 6.3 | 0.0

11. Secondary Outcome: Number of Participants Who Underwent Repeat Ablation Procedures
Description: Number of participants who underwent repeat ablation procedures were reported.
Time Frame: Up to 12 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 246 | 49
Participants | 14 | 3

12. Secondary Outcome: Percentage of Participants With PVs Re-isolation Among All of the Targeted PVs at Repeat Procedure
Description: Percentage of participants with PVs re-isolation among all of the targeted PVs at repeat procedure was reported.
Time Frame: Up to 12 months
Population: The PP set consisted of all enrolled participants who had undergone RF ablation and were treated with the STSF or ST catheters with the VISITAG SURPOINT Module with EPU, and had been treated for the study-related arrhythmia. Here 'N' (number of participants analyzed) signifies the number of participants analyzed in this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 14 | 3
Percentage of Participants | 57.1 | 100

13. Secondary Outcome: Percentage of Participants Requiring New Linear Lesion and/or New Foci Identified During the Repeat Ablation Procedure
Description: Percentage of participants requiring new linear lesion and/or new foci identified during the repeat ablation procedure was reported.
Time Frame: Up to 12 months
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 14 | 3
Percentage of Participants | 64.3 | 66.7

14. Secondary Outcome: Percentage of Participants With 12-Month Single Procedure Success
Description: Percentage of participants with 12-month single procedure success was reported. It is defined as freedom from 1) any repeat procedure for Atrial fibrillation (AF)/Atrial tachycardia (AT)/Atrial flutter (AFL) post index procedure; 2) any class I/III AAD taking during the evaluation period; 3) documented AF/AT/AFL recurrence in evaluation period.
Time Frame: Up to 12 months
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
Number analyzed (Participants) | 236 | 46
Percentage of Participants | 55.5 | 50.0

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: The safety set consisted of all enrolled participants who had undergone insertion of the SMARTTOUCH Surround Flow (STSF) or ST catheter and use of the VISITAG SURPOINT module with external processing unit (EPU).
Arm/Group | VISITAG SURPOINT Module STSF Catheter With EPU | VISITAG SURPOINT Module ST Catheter With EPU
All-Cause Mortality (participants affected / at risk) | 2/261 | 0/49
Serious Adverse Events (participants affected / at risk) | 53/261 | 6/49
Other Adverse Events (participants affected / at risk) | 139/261 | 24/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | VISITAG SURPOINT Module STSF Catheter With EPU (N=261) | VISITAG SURPOINT Module ST Catheter With EPU (N=49)
Cardiac failure (Cardiac disorders) | 4 (4) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 2 (4)
Atrial flutter (Cardiac disorders) | 6 (10) | 2 (2)
Bradycardia (Cardiac disorders) | 4 (4) | 0/0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 2 (2) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 4 (4) | 0 (0)
Pericarditis (Cardiac disorders) | 6 (7) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal angiectasia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 4 (4) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 2 (2)
Electroencephalogram abnormal (Investigations) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 2 (2) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 0 (0)
Peripheral venous disease (Vascular disorders) | 2 (2) | 0 (0)
Death (Nervous system disorders) | 1 (1) | 0 (0)
Cardiac Tamponade/Perforation (Cardiac disorders) | 3 (4) | 0 (0)
Stroke/Cerebrovascular Accident (CVA) (Nervous system disorders) | 1 (1) | 2 (2)
Major Vascular Access Complication / Bleeding (Vascular disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | VISITAG SURPOINT Module STSF Catheter With EPU (N=261) | VISITAG SURPOINT Module ST Catheter With EPU (N=49)
Supraventricular tachycardia (Cardiac disorders) | 12 (12) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 4 (4) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 10 (10) | 2 (2)
Atrial flutter (Cardiac disorders) | 14 (14) | 4 (4)
Atrial tachycardia (Cardiac disorders) | 8 (8) | 0 (0)
Atrioventricular block (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 4 (4) | 2 (2)
Bundle branch block (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 14 (14) | 4 (4)
Pericarditis (Cardiac disorders) | 8 (8) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (6) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 6 (6) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (4) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 6 (6) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 4 (4) | 2 (2)
Intracardiac mass (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Dermoid cyst (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Thyroid mass (Endocrine disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 2 (2)
Visual impairment (Eye disorders) | 2 (2) | 4 (4)
Vitreous floaters (Eye disorders) | 4 (4) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 4 (4) | 0 (0)
Melaena (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Application site laceration (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 4 (4) | 0 (0)
Chest discomfort (General disorders) | 8 (8) | 4 (4)
Chest pain (General disorders) | 31 (34) | 1 (1)
Fatigue (General disorders) | 10 (10) | 2 (2)
Local swelling (General disorders) | 2 (2) | 0 (0)
Oedema (General disorders) | 4 (4) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 6 (6) | 0 (0)
Oedema peripheral (General disorders) | 12 (12) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 2 (2) | 0 (0)
Corona virus infection (Infections and infestations) | 6 (6) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Gingivitis (Infections and infestations) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 2 (2) | 0 (0)
Medical device site infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 8 (12) | 2 (2)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Tooth abscess (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 10 (10) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 10 (10) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Nail avulsion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Scapula fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular access site bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular access site swelling (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
Blood sodium decreased (Investigations) | 0 (0) | 2 (2)
Heart rate increased (Investigations) | 0 (0) | 4 (4)
Weight increased (Investigations) | 0 (0) | 4 (4)
Blood uric acid increased (Investigations) | 2 (2) | 0 (0)
Blood cholesterol increased (Investigations) | 2 (2) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Gout (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 14 (14) | 0 (0)
Headache (Nervous system disorders) | 14 (14) | 0 (0)
Migraine with aura (Nervous system disorders) | 4 (4) | 2 (2)
Presyncope (Nervous system disorders) | 2 (2) | 2 (2)
Sciatica (Nervous system disorders) | 4 (4) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 4 (4)
Vestibular migraine (Nervous system disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2)
Depression (Psychiatric disorders) | 4 (4) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 0 (0)
Dysuria (Renal and urinary disorders) | 4 (6) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (4) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0/40 (0)
Renal pain (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 6 (6) | 0 (0)
Dysuria, Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 (28) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary haemorrhageq (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 4 (4) | 0 (0)
Essential hypertension (Vascular disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 14 (14) | 2 (2)
Haemorrhage (Vascular disorders) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 22 (24) | 2 (2)
Hypotension (Vascular disorders) | 8 (10) | 2 (2)
Labile blood pressure (Vascular disorders) | 2 (2) | 0 (0)
Peripheral venous disease (Vascular disorders) | 2 (2) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT03624881/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT03624881/SAP_001.pdf